CLINICAL TRIAL: NCT04227522
Title: Rucaparib MAintenance After Bevacizumab Maintenance Following Carboplatin Based First Line Chemotherapy in Ovarian Cancer Patients
Acronym: MAMOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NOGGO ov42
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Clear Cell Carcinoma
Keywords: Rucaparib; maintenance therapy; Bevacizumab; Ovarian Cancer; BRCA negative
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Adenocarcinoma, Clear Cell | interventions — rucaparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Rucaparib) (Experimental): Rucaparib treatment (starting dose 600 mg, twice daily) after receiving Bevacizumab for 12 to 15 months. Cycles continue until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria.
  Interventions: Drug: Rucaparib
- Arm B (Placebo) (Placebo Comparator): Placebo treatment after receiving Bevacizumab for 12 to 15 months. Cycles continue until disease progression and/or death, unacceptable adverse event/s, patient and/or investigator decision, other protocol stopping criteria.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Rucaparib — A starting dose of 600 mg Rucaparib is taken twice daily orally by the patients as maintenance after previous maintenance therapy (Bevacizumab) for a period of 12 to 15 months.
  Arms: Arm A (Rucaparib)
Drug: Placebos — Placebo is taken daily orally by the patients as maintenance after previous maintenance therapy (Bevacizumab) for a period of 12 to 15 months.
  Arms: Arm B (Placebo)

SUMMARY:
MAMOC is a multicenter, randomized, placebo controlled, double blind study including BRCA negative patients with histologically confirmed, advanced (FIGO stage IIIA, IIIB, IIIC, or IV of the 2014 FIGO classification) high grade serous or high grade endometrioid (based on local histopathological findings) ovarian cancer, fallopian tube cancer, primary peritoneal cancer and clear cell carcinoma of the ovary in first line therapy.

DETAILED DESCRIPTION:
The main scope of this trial is to determine progression free survival in BRCA negative patients treated with Rucaparib as maintenance therapy vs. Placebo after receiving Bevacizumab for 12 to 15 months.

BRCA negative patients will be stratified according to time point of surgery (adjuvant vs. neoadjuvant), result of surgery (tumor free vs. not tumor free resection), study site and response (complete response (CR) vs. partial response (PR)/SD) and randomized 2:1 to receive either Rucaparib (Arm A) or Placebo (Arm B).

In both of the arms, tumor assessments (CT or MRI) are performed before randomization, and every 6 months thereafter.

During treatment, clinical visits (blood cell counts, detection of toxicity) occur every 4 weeks. Physical examinations will take place every 12 weeks. Safety will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs).

About 30 sites in Germany will participate in this study to recruit 190 BRCA negative patientsin 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18.
3. Patients with histologically confirmed, advanced (FIGO stage IIIA, IIIB, IIIC, or IV of the 2014 FIGO classification) high grade serous or high grade endometrioid (based on local histopathological findings) ovarian cancer, fallopian tube cancer, primary peritoneal cancer and clear cell carcinoma of the ovary in first line therapy.
4. Availability of archival tumor tissue for central next-generation sequencing (NGS) Analysis and no Detection BRCA mutation (BRCAnegative).
5. Treatment with Bevacizumab or respective biosimilar for 12 to 15 months, independent of dosage.
6. Patients who have completed first line platinum-taxane chemotherapy and at least stable disease after treatment with Bevacizumab before randomization.
7. Patients must be randomized at least 3 weeks and no more than 9 weeks after their last dose of Bevacizumab (last dose is the day of the last infusion) and all major toxicities from the previous chemotherapy must have resolved to CTCAE grade 1 or better (except alopecia and peripheral neuropathy).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
9. Patients must have normal organ and bone marrow function:

   1. Hemoglobin ≥ 10.0 g/dL independent of transfusion ≤ 14 days prior to Screening hemoglobin assessment
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109 /L
   3. Platelet count ≥ 100 x 109 /L
   4. Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN); < 2 × ULN if hyperbilirubinemia is due to Gilbert's syndrome
   5. Aspartate aminotransferase /Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤3 x ULN, unless liver metastases are present in which case they must be ≤ 5 x ULN
   6. Serum creatinine ≤ 1.5 x institutional ULN and creatinine clearance > 30 mL/min
   7. Patients not receiving anticoagulant medication who have an International Normalized Ratio (INR) ≤1.5 and an Activated ProThrombin Time (aPTT) ≤1.5 x ULN.
10. Postmenopausal or evidence of non-childbearing status for women of childbearing potential prior to the first dose of study treatment. Female patients of childbearing potential must have a negative serum pregnancy test result ≤3 days prior to administration of the first dose of rucaparib.

Patients are considered to be of childbearing potential unless 1 of the following applies:

1. Considered to be permanently sterile. Permanent sterilization includes hysterectomy, bilateral salpingectomy, and/or bilateral oophorectomy; or
2. Is postmenopausal, defined as no menses for at least 12 months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level consistently in the postmenopausal range (30 milli International Units/milliliter (mIU/mL) or higher) may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy; however, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to confirm a postmenopausal state.

Female patients of reproductive potential must practice highly effective methods (failure rate < 1% per year) of contraception with their partners, if of reproductive potential, during treatment and for 6 months following the last dose of rucaparib or longer if requested by local authorities. Highly effective contraception includes: Ongoing use of progesterone only injectable or implantable contraceptives; Placement of an intrauterine device (IUD) or intrauterine system (IUS); Bilateral tubal occlusion; Sexual abstinence as defined as complete or true abstinence, acceptable only when it is the usual and preferred lifestyle of the patient; periodic abstinence (eg, calendar, symptothermal, post-ovulation methods) is not acceptable; or Sterilization of the male partner, with appropriate post-vasectomy documentation of absence of sperm in ejaculate.

Exclusion Criteria:

1. Non-epithelial origin of the ovary, the fallopian tube or the peritoneum (i.e. germ cell tumors) and Ovarian tumors of low malignant potential (e.g. borderline tumors), or low grade serous ovarian cancer, or low grade endometrioid ovarian cancer, or mucinous carcinoma.
2. Patients with myelodysplastic syndrome/acute myeloid leukemia history.
3. Patients receiving radiotherapy within 6 weeks prior to study treatment.
4. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
5. Previous allogeneic bone marrow transplant.
6. Use of any other PARP-inhibitor in first line therapy.
7. Administration of other simultaneous chemotherapy drugs, any other anti-cancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroidal antiemetics).
8. Clinically significant (e.g. active) cardiovascular disease.
9. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months prior to randomization.
10. History or evidence of hemorrhagic disorders within 6 months prior to randomization.
11. Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).
12. History or evidence for brain metastases or spinal cord compression.
13. History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
14. Significant traumatic injury during 4 weeks prior to randomization.
15. Non-healing wound, active ulcer or bone fracture. Patients with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection are eligible but require 3 weekly wound examinations.
16. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.
17. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.
18. Pregnant or lactating women, women of child-bearing potential who do not agree to the usage of highly effective contraception methods (see inclusion criteria).
19. Participation in another clinical study with an investigational product immediately prior to randomization.
20. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
21. Patients with a known hypersensitivity to Rucaparib or any of the recipients of the product.
22. Known human immunodeficiency virus (HIV) or acquired immunodeficiency Syndrome (AIDS)-related illness, or history of chronic hepatitis B or C.
23. Other active malignancy requiring treatment.
24. Patient who might be dependent on the sponsor, Clinical Research Organization (CRO), site or the investigator.
25. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 Arzneimittelgesetz (AMG).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 48 months
  time from randomization until disease progression or death

SECONDARY OUTCOMES:
Progression free survival 2 (PFS2) | 48 months
  time from randomization to second progression or death
Quality of Life (QoL) 1 | 48 months
  Patients are asked to answer the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30). Responses of questions 1-28 are based on a 4-point scale (1=not at all; 4=Very much), with a higher score indicating a high degree of symptomatology and must therefore be assessed negatively. Responses of questions 29 and 30 are based on a 7-point scale (1=Very poor; 7=Excellent), with a higher score indicating a better global health status.
Quality of Life 2 | 48 months
  Patients are asked to answer the EORTC QoL Questionnaire-Ovarian Cancer (QLQ-OV28). Responses are based on a 4-point scale (1=Not at all; 4=Very much), with a lower score indicating better symptoms.
Quality of Life/ Global health status 3 | 48 months
  Patients are asked to answer the short version of the SF-36 Health Survey (SF-12). The questionnaire contains a total of 12 questions with different response options. For questions 1, 8 and 12 there are 5 (1=excellent, 5=bad), for question 2-3 there are 3 (1=yes, very restricted, 3=no, not restricted at all) and for questions 9-11 there are 6 response options (1= always, 6 = never). Questions 4-7 can be answered with "Yes" or "No".
Quality of Life 4 | 48 months
  Patients are asked to answer the questionnaire Fatigue Symptom Inventory (FSI). Responses are based on a 10 point grading scale (0=not at all tired/ exhausted; 10=completely tired/ exhausted), with a lower score indicating a lower symptomatology of fatigue.
Quality of Life 5 | 48 months
  Patients are asked to answer the Everyday Memory Questionnaire. Responses are based on a 5-point scale (1=occasionally; 5=very often), with a lower score indicating a better performance on memory associated Everyday activities.
Quality of Life 6 | 48 months
  Patients are asked to answer a custom form of the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events developed by the National Cancer Institute (NCI PRO-CTCAE™) Version 1.0. The frequency and strength of symptoms is queried. There are 5 possible answers: "not at all", "a little", "moderate", "quite", "very".
Determination of time to next medical intervention | 48 months
  (e.g. bowel obstruction, Ascites puncture)
Time to next subsequent therapy | 48 months
  e.g. chemotherapy
Number of participants with treatment-related adverse events and/or serious adverse events as assessed by CTCAE v4.03 | 48 months
  AEs/SAEs
Overall survival (OS) | 72 months
  defined as time from Randomization to death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum
Locations (17):
- Germany (17):
  - Universitätsklinikum Aachen, Aachen
  - ANregiomed Frauenklinik Ansbach, Ansbach
  - Helios Klinikum Berlin-Buch, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Kliniken Essen Mitte, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - ViDia Christliche Kliniken Karlsruhe Vincentius-Diakonissen-Kliniken g AG, Karlsruhe
  - Städtisches Krankenhaus Kiel, Kiel
  - ZAGO-Zentrum für ambulante gynäkologische Onkologie, Krefeld
  - Universitätsklinikum Mannheim, Mannheim
  - LMU Klinikum Großhadern, München
  - Universitätsklinikum Münster, Münster
  - CaritasKlinikum Saarbrücken, Saarbrücken
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: Yes
Scienctists may submit a request for scientific use of the data after the first publication. This request shall be examined by the working group.
  After signing an agreement, the anonymous data can be made available to the scientist (password protected).
Supporting Information: Study Protocol, ICF
Time Frame: after first main publication

REFERENCES:
- [Derived] Malhan D, Hesse J, Nelson N, Stankov K, Nguyen J, Aboumanify O, Garmshausen J, Rogmans G, Czogalla B, Gerber J, Koch M, Kupec T, Tome O, Witteler R, Deryal M, Eichbaum M, Sehouli J, Braicu EI, Relogio A. Circadian rhythm disruption by PARP inhibitors correlates with treatment toxicity in patients with ovarian cancer and is a predictor of side effects. EBioMedicine. 2025 Jul;117:105764. doi: 10.1016/j.ebiom.2025.105764. Epub 2025 May 16. PMID 40382284